CLINICAL TRIAL: NCT03310320
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 1b Study to Assess Efficacy and Safety of One Dose Level of Oral AZD0284 Given for Four Weeks, Compared to Placebo, in Patients With Moderate to Severe Plaque Psoriasis
Brief Title: Study to Determine if AZD0284 is Effective and Safe in Treating Plaque Psoriasis
Acronym: DERMIS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study is temporarily suspended due to preclinical findings that are currently under evaluation
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D7800C00003; 2017-002351-29 (EudraCT Number)
Record Dates: First submitted 2017-10-11; First posted 2017-10-16 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Plaque Psoriasis Vulgaris
Keywords: Plaque psoriasis; PASI; BSA; sPGA; P-VAS; IL17A-; CCL20; PK
MeSH Terms: interventions — AZD-0284

STUDY DESIGN:
Intervention Model Description: This is a randomised, double-blind, placebo-controlled, multi-centre, parallel group Phase 1b study in patients with moderate to severe plaque psoriasis. The study is designed to evaluate the pharmacodynamic effects, clinical efficacy and safety of AZD0284 compared with placebo as measured by the relative change from baseline in Psoriasis Area and Severity Index score and biomarkers associated with the mechanism of disease and AZD0284. It comprises 8 clinic visits over approximately 10 weeks including screening visit.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study is double-blind; patients, study site personnel and AZ personnel involved in the evaluation of the data must be kept blinded.
  Packaging and labelling of study drug will be performed in a way that ensures blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo for AZD0284 oral solution
  Interventions: Drug: Placebo
- AZD0284 (Experimental): AZD0284 oral solution 2.5 mg/mL
  Interventions: Drug: AZD0284 oral solution 2.5 mg/mL

INTERVENTIONS:
Drug: AZD0284 oral solution 2.5 mg/mL — AZD0284 oral solution 2.5 mg/mL, 100 mg twice daily for for 4 weeks
  Other Names: AZD0284
  Arms: AZD0284
Drug: Placebo — Placebo for AZD0284 oral solution, twice daily for 4 weeks
  Arms: Placebo

SUMMARY:
The Sponsor is developing the study drug, AZD0284, for the potential treatment of Plaque psoriasis. Psoriasis is a skin condition that causes red, flaky, crusty patches of skin covered with silvery scales. The severity of the disease varies, but in many cases it can have a major impact on their quality of life if not adequately treated.

The purpose of the study is to determine the short term safety, pharmacodynamic and clinical effect of AZD0284 in patients with psoriasis.

DETAILED DESCRIPTION:
This is a randomised, double-blind, placebo-controlled, multi-centre, parallel group Phase 1b study, designed to evaluate the pharmacodynamic effects, clinical efficacy and safety of AZD0284 compared with placebo as measured by the relative change from baseline in Psoriasis Area Severity Index (PASI score), other disease assessments of involved body surface area (BSA), static physicians global assessment score (sPGA), pruritis and biomarkers associated with the mechanism of disease and AZD0284. Disease activity will be assessed throughout the study as will changes in skin biopsy biomarkers. The study population will be comprised of patients with moderate to severe plaque psoriasis as defined by PASI score, BSA and sPGA.

Following completion of screening assessments and meeting all eligibility criteria, patients will be randomised to receive AZD0284 or placebo for 4 weeks of treatment followed by a 4 week follow up period

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent prior to any study specific procedures.
* At least 6 months documented history with a diagnosis of moderate to severe plaque psoriasis as defined by the Psoriasis Area and Severity Index (PASI), psoriasis Body Surface Area (BSA) and static Physician Global Assessment (sPGA).

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the patient at risk because of participation in the study, or influence the results or the patient's ability to participate in the study.
* History and/or presence of tuberculosis, hepatitis, HIV. Other opportunistic infections within 6 months of the study.
* Clinically significant laboratory abnormalities.
* Clinically important abnormalities in rhythm, conduction or morphology of the digital Electrocardiogram (ECG) as considered by the Investigator may interfere with the interpretation of study data.
* Current treatment or treatment for psoriasis with biological therapies within 6 months of study.
* Efficacy and safety failure of biologic therapies targeting the IL-17 and IL12/23 pathway at any time.
* Current treatment or history of treatment for psoriasis with non-biological systemic medications within 4 weeks of Day 1

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Reduction from baseline to the end of treatment, in gene expression level of IL-17A and CCL20 relative to placebo. | 4 weeks
  Reduction from baseline to the end of treatment, in gene expression level of IL-17A and CCL20 relative to placebo.
Percent improvement from baseline to the end of treatment in individual Psoriasis Area and Severity Index (PASI) compared to placebo | 4 weeks
  Change (percent improvement) in Psoriasis Area and Severity Index score(PASI) compared to placebo

SECONDARY OUTCOMES:
Proportion of patients achieving 75 % reduction from baseline in PASI score, i.e. PASI 75, at week 4 | 4 weeks
  Percent patients acheiving a 75% reduction in PASI score
Proportion of patients achieving 50 % reduction from baseline in PASI score, i.e. PASI 50, at week 4 | 4 weeks
  Percent patients acheiving a 50% reduction in PASI score
Reduction in static physician's global assessment (sPGA) score from baseline at week4 | 4 weeks
  The change in the Static physician's global assessment (sPGA) score will be assessed
Percent improvement from baseline in involved body surface area (BSA) at week 4 | 4 weeks
  The percent change in the involved body surface area (BSA) will be assessed
Reduction in the pruritus visual analogue scale (pVAS) score from baseline, at week 4 | 4 weeks
  The reduction in the pruritus visual analogue scale (pVAS) score as determined by the patient will be assessed
Cmax : maximum observed plasma concentration | 4 weeks
  Maximum observed plasma concentration (Cmax) will be assessed
tmax time to reach Cmax | 4 weeks
  The time to reach the maximum observed plasma concentration (Cmax) will be assessed
Cmin minimum observed plasma concentration | 4 weeks
  The minimum observed plasma concentration (Cmin) will be assessed
AE(s) and SAE(s) | Approximately 8 weeks throughout the study
  Safety evaluation will include the assessment of adverse and serious adverse events over the course of the study

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Psallidas, Phd, Study Director — AstraZeneca R&D, Gothenburg, Sweden
Locations (4):
- Denmark (4):
  - Research Site, Aarhus C
  - Research Site, Copenhagen
  - Research Site, Hellerup
  - Research Site, Odense

IPD SHARING:
Plan to Share IPD: No